CLINICAL TRIAL: NCT02315261
Title: Effectiveness of Epidural Anesthesia for Thoracic and Abdominal Surgery in Siriraj Hospital
Brief Title: Effectiveness of Epidural Anesthesia for Thoracic and Abdominal Surgery
Status: Completed | Type: Observational
Sponsor: Siriraj Hospital (Other)
Responsible Party: Principal Investigator, Mingkwan Wongyingsinn, MD, Assistant professor, Doctor, Siriraj Hospital
Other Study IDs: SIRB004
Record Dates: First submitted 2014-12-04; First posted 2014-12-11 (Estimated); Results first posted 2018-11-13 (Actual); Last update posted 2018-11-13 (Actual); Status verified 2018-04

CONDITIONS: Analgesia Disorder; Anesthetic Complication Epidural; Adverse Reaction to Epidural Anesthesia
Keywords: Epidural analgesia; Pain score
MeSH Terms: interventions — Analgesia, Epidural

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Elective Thoracic and Abdominal Surgery Patients — This is an observational audit, reviewing the implementation of a standard care practice and requiring de-identified data collection in Elective Thoracic and Abdominal Surgery Patients only. All collected data will be that which is routinely part of normal clinical practice. The Research staff will systematically collect data on each patient. Some information can be obtained from the medical record, intraoperative anesthetic record, acute pain service record, etc whereas other information has to be obtained from direct observation at the bedside.
  Other Names: Epidural Analgesia

SUMMARY:
This study aims to evaluate the effectiveness of the epidural analgesia in patients having elective thoracic and abdominal surgery under general anesthesia combined with epidural analgesia in Siriraj Hospital.

DETAILED DESCRIPTION:
Epidural analgesia is the recommended perioperative analgesia in patients having major surgery in order to significantly reduced pain scores, minimize patient distress and can accelerate postoperative recovery especially with the major operation This technique has been reported to provide better pain control and less postoperative fatigue compared with patients receiving general anesthesia alone.Additionally, it is recommended in patients having major surgery to allow patients to mobilize quickly and have effective mobilization.This technique has been shown to be highly efficient at preventing postoperative ileus and various complications. Moreover, epidural analgesic technique is demonstrated to be safer and have fewer side effects than using intravenous opioids alone.

However, the epidural technique is not universally successful and the number of patients experiencing inadequate analgesia with this technique is approximately 12-32%. The failure of epidural analgesia is still a frequent clinical problem and needs active management including a new block or other analgesic medication in order to rescue postoperative pain. Previous study showed that the incidence of patients having epidural analgesia with postoperative moderate pain was 20.9% and that with severe pain was 7.8%. In Siriraj Hospital, recent study showed that 19.6% of patients having elective upper abdominal surgery under general anesthesia combined with epidural analgesia reported severe first pain scores in post anesthetic care unit.27 As a result of severe pain, patients needed a number of intervention and management from acute pain service, and finally spent longer time in post anesthetic care unit.

Inadequate pain control in patients receiving epidural analgesia frequently occurred in clinical practice but the number of the success rate or the failure rate have not been reported in our hospital. This study aims to evaluate the effectiveness of the epidural analgesia in patients having elective thoracic and abdominal surgery under general anesthesia combined with epidural analgesia in Siriraj Hospital.

ELIGIBILITY:
Inclusion Criteria:

* patients aged more than 18 years old scheduled to have thoracic or abdominal surgery under general anesthesia combined with epidural analgesia in Siriraj hospital

Exclusion Criteria:

* inability to communicate or inform pain score
* cesarean section or labor analgesia
* additional analgesic techniques (spinal analgesia, paravertebral nerve block, intercostal block, transversus abdominis plane block, rectus sheath block, ilioinguinal block, iliohypogastric block
* emergency surgery
* fail epidural block after test dose of local anesthetics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients scheduled to have thoracic or abdominal surgery under general anesthesia combined with epidural analgesia in Siriraj hospital
Sampling Method: Probability Sample
Enrollment: 364 (Actual)
Dates: Start 2014-12; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mingkwan Wongyingsinn, MD, MSc, Principal Investigator — Siriraj Hospital
Locations (1):
- Siriraj Hospital, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wongyingsinn M, Anuwongjaroen A. Effectiveness of Postoperative Epidural Analgesia for Thoracic and Abdominal Surgery in Siriraj Hospital. J Med Assoc Thai. 2016 May;99(5):531-8. PMID 27501608

RESULTS

PARTICIPANT FLOW:
Groups:
- Epidural Group: Patients age > 18 years old scheduled to have thoracic or abdominal surgery under general anesthesia combined with epidural analgesia in Siriraj hospital
Period: Overall Study
Arm/Group | Epidural Group
Started | 364
Completed | 364
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Epidural Group
Number analyzed (Participants) | 364
Age, Continuous [Mean (Standard Deviation); unit: years] | 59 (13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 122
  Male | 242
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 23.9 (5.1)
ASA physical classification [Count of Participants; unit: Participants] — The ASA physical status classification system is a system for assessing the fitness of patients before surgery. In 1963 the American Society of Anesthesiologists (ASA) adopted this category physical status classification system as
  ASA physical status I: Healthy person. ASA physical status II: Mild systemic disease. ASA physical status III: Severe systemic disease. ASA physical status IV: Severe systemic disease that is a constant threat to life.
  Participants
    ASA physical status I | 53
    ASA physical status II | 215
    ASA physical status III | 94
    ASA physical status IV | 2
Surgical site [Count of Participants; unit: Participants]
  Thoracic | 36
  Upper abdomen | 131
  Lower abdomen | 192
  Whole abdomen | 5
Duration of surgery [Mean (Standard Deviation); unit: minutes] | 192 (85)

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Reporting Postoperative Verbal Rating Scale Pain at Rest More Than 7
Description: Verbal Rating Scale Pain will routinely be assessed at postoperative 24 hours by the ward nurse.
  Minimum and maximum scores possible are 0 and 10. The higher values represent patients having more pain. Severe pain is defined as Verbal Rating Scale pain at rest more than 7.
Time Frame: at postoperative 24 hours
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Group
Number analyzed (Participants) | 364
Participants | 89

2. Secondary Outcome: Number of Patients Requiring Rescue Analgesic Medication
Description: Number of patients requiring at least one rescue analgesic medication including epidural catheter, oral and intravenous route after the operation
Time Frame: during the period of retaining of epidural catheter up to 3 days after operation
Measure: Count of Participants; unit: Participants
Arm/Group | Epidural Group
Number analyzed (Participants) | 364
Participants | 50

3. Secondary Outcome: Duration Retaining Epidural Catheter
Description: Duration retaining epidural catheter in hospital
Time Frame: the period of retaining of epidural catheter up to 3 days after operation
Measure: Mean (95% Confidence Interval); unit: hours
Arm/Group | Epidural Group
Number analyzed (Participants) | 364
hours | 55.8 [53.9 to 57.6]

4. Secondary Outcome: All Adverse Effects and Postoperative Complications.
Description: All Adverse Effects and Postoperative Complications included the number of patients having postoperative nausea and vomiting; hypotension; accidental dural puncture and post-dural puncture headache.
Time Frame: the period of retaining of epidural catheter up to 3 days after operation
Measure: Number; unit: participants
Arm/Group | Epidural Group
Number analyzed (Participants) | 364
participants
  Postoperative nausea and vomiting | 100
  Hypotension | 28
  Accidental dural puncture | 5
  Post-dural puncture headache | 3

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Epidural Group
All-Cause Mortality (participants affected / at risk) | 0/364
Serious Adverse Events (participants affected / at risk) | 42/364
Other Adverse Events (participants affected / at risk) | 213/364
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Epidural Group (N=364)
Hypotension (Cardiac disorders) | 28
Motor weakness (Nervous system disorders) | 9
Dural puncture (Injury, poisoning and procedural complications) | 5
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Epidural Group (N=364)
Postoperative nausea and vomitting (Injury, poisoning and procedural complications) | 100
Pruritus (Injury, poisoning and procedural complications) | 109
Urinary retention (Injury, poisoning and procedural complications) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No